CLINICAL TRIAL: NCT02010905
Title: Right Ventricular Dysfunction in Tetralogy of Fallot: Inhibition of the Renin-angiotensin-aldosterone System
Acronym: Redefine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: The Interuniversity Cardiology Institute of the Netherlands (Other Government)
Responsible Party: Principal Investigator, Berto J Bouma, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL44943.018.13
Record Dates: First submitted 2013-12-06; First posted 2013-12-13 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Tetralogy of Fallot; Heart Defects, Congenital; Ventricular Dysfunction, Right
Keywords: Losartan
MeSH Terms: conditions — Tetralogy of Fallot; Heart Defects, Congenital; Ventricular Dysfunction, Right | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Losartan 150mg daily (Active Comparator): Losartan: white film-coated biconvex tablet (50mg) with a diameter of 8mm. One time daily three tablets.
  Interventions: Drug: Losartan
- Placebo 150mg daily (Placebo Comparator): Placebo: white film-coated biconvex tablet (50mg) with a diameter of 8mm. One time daily three tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan
  Arms: Losartan 150mg daily
Drug: Placebo
  Arms: Placebo 150mg daily

SUMMARY:
Rationale: The prevalence of adult patients with congenital heart disease (CHD) has steadily increased over the last decades, due to the advances in cardiac surgery. A large number of these patients cope with right ventricular (RV) volume or pressure overload, largely caused by residual lesions after cardiac surgery in childhood. Previous RV overload due to pulmonary regurgitation in Tetralogy of Fallot (TOF) can lead to RV dysfunction. These findings warrant close surveillance of RV function, and adequate and evidence-based pharmacological therapy to reduce both morbidity and mortality in this young patient group. The renin-angiotensin-aldosterone system (RAAS) is activated in patients with ventricular failure, irrespective of the effected (left or right) ventricle. Angiotensin converting enzyme (ACE) inhibitors and angiotensin II receptor blockers (ARB's) are drugs which act as inhibitors of RAAS. Previously, large trials have demonstrated the beneficial effect of angiotensin converting enzyme (ACE) inhibitors on morbidity and mortality in patients with acquired left ventricular (LV) dysfunction. ARB's have a similar effect as ACE inhibitors in patients with acquired LV dysfunction but discontinuation because of side effects such as cough is less frequent. In TOF patients with RV overload due to pulmonary regurgitation, pulmonary valve replacement leads to a decrease in RV size and pulmonary regurgitation. Current guidelines advise empiric use of RAAS inhibitors for right ventricular dysfunction in adult patients with congenital heart disease. However, the actual effect of RAAS inhibition on right ventricular dysfunction in adult TOF patients without severe valvular lesions has not been sufficiently investigated. Therefore, we set-up the proposed study, and hypothesize that ARB's have a beneficial effect on RV ejection fraction in adult TOF patients with RV dysfunction without severe valvular lesions.

Objective: to improve RV ejection fraction in adult TOF patients with RV dysfunction without severe valvular lesions.

Study design: a prospective, multicenter, double-blind, randomized, placebo-controlled trial. Follow up two years Study population: adult patients with Tetralogy of Fallot with right ventricular dysfunction, defined as right ventricular ejection fraction < 50% and without severe valvular lesions Intervention: patients are randomized to receive either losartan 150 mg once daily, or placebo in the same regimen. Main study parameters/endpoints: the primary endpoint is difference in change in RV ejection fraction, determined by cardiovascular magnetic resonance imaging (CMR), between the treatment and the control group at two years follow-up.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All investigations, except blood analysis, are non-invasive and free of risk. The burden for the patients mainly consists of the time that is consumed by the visits to the clinic. At these visits time will be consumed by: history taking and physical investigation (15 minutes); quality of life score (15 minutes); laboratory tests (6 times venopuncture, total amount of blood withdrawn approximately 90ml). Cardiopulmonary exercise testing (1hour), echocardiography (15 minutes) and CMR (45 minutes) are part of regular medical care. Adverse effects from losartan are usually limited and consist of dizziness due to hypotension, renal impairment, hyperkalemia and liver impairment. We expect no change or an increase in RV function in the intervention group compared to the control group over the two-year follow up period, which would be a great benefit for this young study population.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria: adult age and mentally competent; and Tetralogy of Fallot; and right ventricular dysfunction, defined as right ventricular ejection fraction 50% or lower as measured by Cardiovascular Magnetic Resonance Imaging (CMR). Not more than moderate tricuspid or pulmonary regurgitation or more than moderate pulmonary stenosis as measured by CMR or echocardiography.

Exclusion Criteria:

* Incapable of giving informed consent
* Hypersensitivity to losartan or any of its help substances
* Contraindications for CMR
* Previous or current angioedema whether or not in relation to the use of an ACE inhibitor or ARB
* Known bilateral renal artery stenosis
* Current symptomatic hypotension
* Estimated glomerular filtration rate of 30 ml/min or lower
* Plasma potassium level of 5,5 mmol/L or higher
* Moderate to severe liver disease: Child Pugh class B or C
* Raised plasma transaminases level more than three times upper normal limit
* Current treatment of hypertension with an ACE-inhibitor or ARB, which cannot be discontinued
* Current treatment with potassium chloride, trimethoprim, tacrolimus or cyclosporine which cannot be discontinued
* Pregnant or nursing women
* Desire to have children within the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-12; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Right ventricular ejection fraction | two years
  RV EF is measured by means of cardiovascular magnetic resonance imaging (CMR)

SECONDARY OUTCOMES:
RV volumes (CMR) | two years
pulmonary regurgitation (CMR and echocardiography) | two years
aortic root diameter (CMR and echocardiography) | two years
echocardiographic parameters for RV and LV function | one year and two years
maximal exercise capacity (VO2 max) | two years
hospitalization for heart failure | two years
the prevalence of (supra) ventricular arrhythmias | within two years
the serum ntproBNP levels | one year and two years
NYHA class | two years
Quality of life (SF 36 and SQUASH) | two years
death | two years
RV mass (CMR) | two years
LV EF (CMR) | two years
LV volumes (CMR) | two years
LV mass (CMR) | two years
serum Galectin-3 levels | two years
circulating microRNA's | two years

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (6):
  - Academic Medical Center, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Leids Universitair Medisch Centrum, Leiden
  - St Antonius ziekenhuis, Nieuwegein
  - St Radboud Universitair Medisch Centrum, Nijmegen
  - Universitair Medisch Centrum Utrecht, Utrecht

REFERENCES:
- [Derived] Bokma JP, Winter MM, van Dijk AP, Vliegen HW, van Melle JP, Meijboom FJ, Post MC, Berbee JK, Boekholdt SM, Groenink M, Zwinderman AH, Mulder BJM, Bouma BJ. Effect of Losartan on Right Ventricular Dysfunction: Results From the Double-Blind, Randomized REDEFINE Trial (Right Ventricular Dysfunction in Tetralogy of Fallot: Inhibition of the Renin-Angiotensin-Aldosterone System) in Adults With Repaired Tetralogy of Fallot. Circulation. 2018 Apr 3;137(14):1463-1471. doi: 10.1161/CIRCULATIONAHA.117.031438. Epub 2017 Dec 8. PMID 29222139